CLINICAL TRIAL: NCT05115266
Title: Efficacy of Animal-assisted Therapy in Patients With Borderline Personality Disorder and Addictions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Miguel Monfort Montolio (Other)
Responsible Party: Sponsor-Investigator, Miguel Monfort Montolio, Miguel Monfort Montolio, member of the TXP research group at Cardenal Herrera University, Cardenal Herrera University
Organization: Cardenal Herrera University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAT BPD&A
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Diagnosis, Dual (Psychiatry)
Keywords: Animal-assisted therapy; Borderline personality disorder; substance abuse; Dual pathology; Residential treatment
MeSH Terms: conditions — Disease; Borderline Personality Disorder; Substance-Related Disorders | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (EG) (Experimental): Receive animal-assisted therapy and usual treatment (ATT)
  Interventions: Behavioral: Animal-assisted therapy (AAT
- Control group (Active Comparator): Receive usual treatment
  Interventions: Behavioral: Usual treatment

INTERVENTIONS:
Behavioral: Animal-assisted therapy (AAT — The activity program consists of 10 sessions with a duration of about 60 minutes. During the 10 sessions the animal is presented, in this case a dog. They caress it, dress it, educate it ...
  Other Names: ATT
  Arms: Experimental group (EG)
Behavioral: Usual treatment — receive usual treatment (group activities)
  Arms: Control group

SUMMARY:
Animal-assisted therapy (AAT) is a complementary intervention of therapy that has shown positive results in the treatment of various pathologies. This study assesses the viability of the implementation and the effectiveness of an AAT program in patients diagnosed with borderline personality disorder and substance abuse disorder.

Our hypotheses are that participation in the TAA program will reduce negative symptoms, improve the quality of life of people with dual pathology, whose mental illness is schizophrenia, and increase adherence to treatment for people with dual pathology, whose mental disorder it's schizophrenia.

DETAILED DESCRIPTION:
Animal assisted therapy (AAT) is a complementary intervention to therapy that presents positive results in the treatment of different pathologies. The study assesses the implementation and effectiveness of a TAA program in patients diagnosed with borderline personality disorder and substance abuse disorder.

ELIGIBILITY:
Inclusion Criteria:

* Meeting DSM-5 criteria for substance abuse disorder and the presence of borderline personality disorder.
* Voluntary participant in the study and having signed the informed consent

Exclusion Criteria:

* Patients whose functioning could be altered by factors not specifically related to addictive pathology or mental disorder (severe cognitive impairment, intellectual deficiency or language barrier)
* Animal-specific phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The Life Skills Profile questionnaire (LSP) | Change from Life Skills at 3-6-9 months (12 minutes)
  This questionnaire evaluates aspects of functioning that affect daily activities and the adaptation of people with mental illnesses in the community. It contains 39 items that are grouped into self-care, social-interpersonal behaviour, communication-social contact, non-personal social behavior and autonomous life
Barrat impulsiveness scale (BIS-11) | Change from impulsiveness at 3-6-9 months (12 minutes)
  This instrument is composed of 30 items distributed into three sub-scales: nonplanning, motor and attentional. The total impulsiveness score was also obtained
Calgary Depresión Scale for Schizophrenia (CDSS) | Change from Depresión at 3-6-9 months (12 minutes)
  The questionnaire is a structured instrument, administered by a clinician in a hetero-applied way for the adult population, with an approximate administration time of between 10 and 30 minutes, and covers the therapeutic area related to the symptoms of depressive disorders.
Rosenberg Self-Esteem Scale | Change from self-esteem at 3-6-9 months (12 minutes)
  The questionnaire consists of 10 statements of the feelings that the person has about himself. Five of the statements are addressed positively (items 1, 2, 4, 6 and 7) and 5 negatively (items 3, 5, 8, 9 and 10).
Positive and negative symptom scale (PANSS) | Change from Positive and negative symptom at 3-6-9 months (12 minutes)
  It is a semi-structured and hetero-applied questionnaire for the adult population. The application time is between 30-60 minutes and evaluates the positive and negative symptoms of schizophrenia and other psychotic disorders